CLINICAL TRIAL: NCT07018700
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter, Clinical Trial With Extension Period to Evaluate the Efficacy and Safety of Xeomin® Injections for the Prevention of Episodic Migraine
Brief Title: A Clinical Trial to Evaluate Efficacy and Safety of Xeomin® Injections for Preventing Episodic Migraine
Acronym: MINT-E
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merz Therapeutics GmbH (Industry)
Responsible Party: Sponsor
Organization: Merz Pharmaceuticals GmbH (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M602011085; 2024-515715-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-04; First posted 2025-06-12 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Episodic Migraine
MeSH Terms: interventions — incobotulinumtoxinA; Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Xeomin Dose A (Experimental): Placebo-controlled period + extension period: Xeomin injections at pericranial and cervical points (dose A)
  Interventions: Drug: Xeomin
- Xeomin Dose B (Experimental): Placebo-controlled period + extension period: Xeomin injections at pericranial and cervical point (dose B)
  Interventions: Drug: Xeomin
- Placebo (Placebo Comparator): Placebo-controlled period: Placebo injections at pericranial and cervical points.
  Extension period: Xeomin injections at pericranial and cervical points (dose A)
  Interventions: Drug: Xeomin; Drug: Placebo

INTERVENTIONS:
Drug: Xeomin — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl)
  Other Names: IncobotulinumtoxinA; NT 201; Botulinum toxin type A (150 kiloDalton), free from complexing proteins
Drug: Placebo — Solution for injection prepared by reconstitution of powder with 0.9% Sodium Chloride (NaCl)
  Arms: Placebo

SUMMARY:
In this clinical trial, participants with episodic migraine will receive injections with Xeomin or Placebo into muscles of the head and neck. The purpose is to measure the change in monthly migraine days with Xeomin injections compared to Placebo injections.

Trial details include:

* Trial duration: 52 to 55 weeks;

  * Screening period: 4 to 5 weeks;
  * Treatment duration: 4 treatments, each about 12 weeks apart; and
* Visit frequency: about every 4 weeks, 14 visits in total. The first and last visit and the 4 treatment visits are on-site, the other 8 visits are remote by phone / video call.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a diagnosis of EM with or without aura according to current International Classification of Headache Disorders (Edition 3 and Edition 4 alpha) criteria for ≥ 12 months and is able to distinguish migraine headaches from all other types of headaches;
* Participant age < 50 years at the time of migraine onset;
* Participant meeting the following headache and migraine day criteria in each of the 3 months prior to screening: history of ≤ 14 headache days per month and history of 6 to 14 migraine days per month; and
* During the last 28 days of the screening period, participant experiencing: ≤ 14 headache days and 6 to 14 migraine days that qualify as such per the headache diary.

Exclusion Criteria:

* Diagnosis of chronic migraine;
* Diagnosis of other primary headache types, except tension-type headache, which is permitted;
* Diagnosis of aura without headache, migraine with brainstem aura, hemicrania continua, hypnic headache, hemiplegic migraine, retinal migraine, persistent aura without infarction, migraine aura-triggered seizure, or previous migrainous infarction;
* Diagnosis of secondary headache types, except medication overuse headache, which is permitted;
* Currently taking > 1 prescribed drug for the preventive treatment of migraine;
* Discontinuation of anti-calcitonin gene-related peptide (CGRP) / anti-CGRP receptor monoclonal antibody treatment less than 5 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 990 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Change in monthly migraine days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose A | Baseline to month 6

SECONDARY OUTCOMES:
Change in monthly migraine days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose B | Baseline to month 6
Change in monthly headache days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose A | Baseline to month 6
Change in monthly headache days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose B | Baseline to month 6
Change in monthly acute migraine medication days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose A | Baseline to month 6
Change in monthly acute migraine medication days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection) - Dose B | Baseline to month 6
Change in frequency of migraine days from baseline (baseline monthly migraine days divided by 2) to two-week end-of-cycle periods (weeks 11 and 12 of Cycle 1 to 4) | Baseline up to 12 months
Percentage of participants who reported at least a 50% reduction in mean monthly migraine days from baseline (28 days before baseline visit) to Month 6 (weeks 21 to 24 after first injection | Baseline to month 6
Incidence of treatment-emergent adverse events (TEAEs) related to treatment as assessed by the investigator in the placebo-controlled period | Month 6

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz Therapeutics
Locations (87):
- United States (39):
  - Arizona Neuroscience Research, Merz Investigational Site #0010521, Phoenix, Arizona
  - Baptist Health Medical Center, Merz Investigational Site #0010520, Little Rock, Arkansas
  - Chemidox Clinical Trials Inc, Merz Investigational Site #0010488, Lancaster, California
  - Clinical Research Institute, Merz Investigational Site #0010487, Los Angeles, California
  - Clinical Trials Management Services, Merz Investigational Site #0010526, Thousand Oaks, California
  - BNL Health Inc., Merz Investigational Site #0010489, Torrance, California
  - Hasbani Neurology, Merz Investigational Site #0010509, New Haven, Connecticut
  - New England Institute Neurology and Headache, Merz Investigational Site #0010441, Stamford, Connecticut
  - Northwest Florida Clinical Research Group, Merz Investigational Site #0010286, Gulf Breeze, Florida
  - Nexus Clinical Research Center, Merz Investigational Site #0010514, Homestead, Florida
  - Jacksonville Center for Clinical Research, Merz Investigational Site #0010515, Jacksonville, Florida
  - Clinical Research of Central Florida, Merz Investigational Site #0010532, Lakeland, Florida
  - American Research Institute, Merz Investigational Site #0010492, Miami, Florida
  - Premiere Research Institute at Palm Beach Neurology, Merz Investigational Site #0010499, West Palm Beach, Florida
  - Accel Research - NeuroStudies, Merz Investigational Site #0010523, Decatur, Georgia
  - Hawaii Pacific Neuroscience, Merz Investigational Site #0010510, Honolulu, Hawaii
  - Kansas Institute of Research,, Merz Investigational Site #0010495, Overland Park, Kansas
  - Crescent City Headache and Neurology Center, Merz Investigational Site #0010517, Chalmette, Louisiana
  - DelRicht Clinical Research,, Merz Investigational Site #0010518, New Orleans, Louisiana
  - Sinai Hospital of Baltimore, Merz Investigational Site #0010505, Baltimore, Maryland
  - MedVadis Research, Merz Investigational Site #0010524, Waltham, Massachusetts
  - Mass Institute of Clinical Research, Merz Investigational Site #0010506, Westborough, Massachusetts
  - Vida Clinical Studies, Merz Investigational Site #0010498, Dearborn Heights, Michigan
  - Quest Research Institute, Merz Investigational Site #0010484, Farmington Hills, Michigan
  - StudyMetrix Research, Merz Investigational Site #0010530, City of Saint Peters, Missouri
  - Quality Clinical Research, Merz Investigational Site #0010522, Omaha, Nebraska
  - Dent Neurosciences Research Center, Merz Investigational Site #0010486, Amherst, New York
  - Integrative Clinical Trials, Merz Investigational Site #0010496, Brooklyn, New York
  - New York Neurology Associates, Merz Investigational Site #0010500, New York, New York
  - True North Neurology, Merz Investigational Site #0010508, Port Jefferson Station, New York
  - Rochester Clinical Research, Merz Investigational Site #0010512, Rochester, New York
  - Upstate Clinical Research Associates, Merz Investigational Site #0010485, Williamsville, New York
  - Dayton Center for Neurological Disorders, Merz Investigational Site #0010531, Centerville, Ohio
  - Headache Center of Hope, Merz Investigational Site #0010528, Cincinnati, Ohio
  - Tekton Research, Merz Investigational Site #0010494, Edmond, Oklahoma
  - Coastal Neurology, Merz Investigational Site #0010503, Port Royal, South Carolina
  - Alina Clinical Trials, Merz Investigational Site #0010511, Dallas, Texas
  - Lone Star Neurology, Merz Investigational Site #0010497, Frisco, Texas
  - Gundersen Health System, Merz Investigational Site #0010507, La Crosse, Wisconsin
- Klinikum Klagenfurt Am Wörthersee, Merz Investigational Site #0430042, Klagenfurt, Austria
- Rigshospitalet-Glostrup, Merz Investigational Site #0450006, Glostrup Municipality, Denmark
- France (2):
  - CHU Clermont Ferrand, Merz Investigational Site #0330026, Clermont-Ferrand
  - CHU Nantes, Merz Investigational Site #0330068, Nantes
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Merz Investigational Site #0490398, Berlin
  - Kopfschmerzzentrum Frankfurt, Merz Investigational Site #0490394, Frankfurt
  - Universitätsmedizin Greifswald, Merz Investigational Site #0490397, Greifswald
  - Vitos Orthopädische Klinik Kassel, Merz Investigational Site #0490396, Kassel
  - Schmerzklinik Kiel GmbH, Merz Investigational Site #0490395, Kiel
- Italy (5):
  - Azienda Ospedaliera Universitaria Careggi, Merz Investigational Site #0390023, Florence
  - Ospedale San Raffaele, Merz Investigational Site #0390027, Milan
  - Istituto Auxologico Italiano, Merz Investigational Site #0390024, Milan
  - Fondazione Istituto Neurologico Nazionale Casimiro Mondino, Merz Investigational Site #0390025, Pavia
  - IRCCS San Raffaele Roma, Merz Investigational Site #0390026, Roma
- Poland (18):
  - Centrum Medyczne Neuromed, Merz Investigational Site #0480117, Bydgoszcz
  - AthleticoMed, Merz Investigational Site #0480127, Bydgoszcz
  - ETG Debica, Merz Investigational Site #0480121, Dębica
  - Centrum Medyczne Pratia Gdynia, Merz Investigational Site #0480126, Gdynia
  - Silmedic Sp. z o.o., Merz Investigational Site #0480115, Katowice
  - Jan Banach Research Spot, Merz Investigational Site #0480059, Krakow
  - Pratia MCM, Merz Investigational Site #0480087, Krakow
  - FutureMeds, Merz Investigational Site #0480125, Krakow
  - Krakowska Akademia Neurologii, Merz Investigational Site #0480031, Krakow
  - Neurocor, Merz Investigational Site #0480119, Krakow
  - ETG Lublin, Merz Investigational Site #0480118, Lublin
  - Indywidualna Praktyka Lekarska Dr hab. Med. Anna Szczepańska-Szerej, Merz Investigational Site #0480096, Lublin
  - Instytut Zdrowia dr Boczarska-Jedynak, Merz Investigational Site #0480103, Oświęcim
  - Solumed Centrum Medyczne, Merz Investigational Site #0480122, Poznan
  - ETG Neuroscience, Merz Investigational Site #0480116, Warsaw
  - MIGRE Polskie Centrum Leczenia Migreny, Merz Investigational Site #0480124, Wroclaw
  - Futuremeds, Merz Investigational Site #0480123, Wroclaw
  - ETG Zamosc, Merz Investigational Site #0480120, Zamość
- Slovakia (3):
  - MUDr. Beáta Dupejová, neurologická ambulancia, Merz Investigational Site #4210002, Banská Bystrica
  - KONZÍLIUM, Merz Investigational Site #4210011, Dubnica nad Váhom
  - NEURES, Merz Investigational Site #4210006, Krompachy
- Spain (13):
  - Hospital Clinic de Barcelona-Hospital Plato, Merz Investigational Site #0340047, Barcelona
  - Hospital Universitari Vall d'Hebron, Merz Investigational Site #0340006, Barcelona
  - Hospital Universitario 12 de Octubre, Merz Investigational Site #0340055, Madrid
  - Hospital Universitario La Paz, Merz Investigational Site #0340007, Madrid
  - Campus Blua Sanitas Valdebebas Hospital, Merz Investigational Site #0340057, Madrid
  - Hospital Regional Universitario de Malaga, Merz Investigational Site #0340050, Málaga
  - Hospital Universitario Virgen de la Victoria, Merz Investigational Site #0340056, Málaga
  - Hospital Vithas Malaga, Merz Investigational Site #0340054, Málaga
  - Hospital Universitario Virgen del Rocio, Merz Investigational Site #0340046, Seville
  - Consorci Sanitari de Terrassa, Merz Investigational Site #0340051, Terrassa
  - Hospital Universitari i Politecnic La Fe de Valencia, Merz Investigational Site #0340049, Valencia
  - Complejo Hospitalario Universitario de Vigo, Merz Investigational Site #0340052, Vigo
  - Hospital Viamed Montecanal, Merz Investigational Site #0340053, Zaragoza

IPD SHARING:
Plan to Share IPD: No